CLINICAL TRIAL: NCT06530043
Title: Effects of Senobi Exercises Versus Jacobsons Muscular Relaxation Exercises on Pulmonary Functions, Dyspnea, and Sleep Quality in Chronic Obstructive Pulmonary Disease
Brief Title: Comparing Senobi and Jacobsons Exercises in COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0374
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Jacobsons Muscular relaxation exercises, Senobi exercises
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Senobi exercises (Experimental): * Group A had undergone Senobi exercises training, scheduled three times weekly over 8 weeks, for individuals with COPD the duration and time interval time for Senobi exercises can vary depending on their overall health, fitness level, and tolerance.
  * The session began with the comfortable sitting of participants with slow inhalation, filling the lungs for a count of 4-5 seconds and holding the breath for 2-3 seconds.
  * In the second step exhale slowly through the mouth, emptying the lungs for a count of 4-5 seconds, and hold the breath for 2-3 seconds.
  * The session started with a shorter session (3-5 minutes) and increased gradually as participants built up endurance with a breathing rate of 4-6 breaths per minute.
  * The cycle of Senobi exercises was repeated for 5-10 minutes and 2-3 times a day.
  Interventions: Other: Senobi exercises
- Jacobsons Muscular relaxation exercises (Experimental): * Group B engaged in a Jacobsons Muscular relaxation exercises plan, following the same frequency and duration as the Senobi exercise program-three sessions per week for 8 weeks.
  * The session started by tensing the muscles in the toes and then moving up the body tensing and relaxing each muscle group in turn (feet and toes, calves, thighs, hips, lower back, upper back, shoulders, arms, hands, neck, and head) and hold it for 5-7 seconds and released it for 5-7 seconds.
  * Repeat the cycle 2-3 times per day with deep breaths between each cycle.
  * The session started with a shorter session (3-5 minutes) and increased gradually as participants built up endurance with a breathing rate of 4-6 breaths per minute.
  Interventions: Other: Jacobsons Muscular relaxation exercises

INTERVENTIONS:
Other: Senobi exercises — Senobi exercise began with the comfortable sitting of participants with slow inhalation, filling the lungs for a count of 4-5 seconds and holding the breath for 2-3 seconds.
  Arms: Senobi exercises
Other: Jacobsons Muscular relaxation exercises — Jacobsons Muscular relaxation exercises started by tensing the muscles in the toes and then moving up the body tensing and relaxing each muscle group in turn (feet and toes, calves, thighs, hips, lower back, upper back, shoulders, arms, hands, neck, and head) and hold it for 5-7 seconds and released it for 5-7 seconds.
  Arms: Jacobsons Muscular relaxation exercises

SUMMARY:
The study aims to evaluate the effects of Senobi versus Jacobsons muscular relaxation exercises on pulmonary functions, dyspnea, and sleep quality in chronic obstructive pulmonary disease. The study design will be a randomized clinical trial. The study will be completed in 10 months after the approval of the synopsis from the Ethical Committee of RCRS and AHS. A non-probability convenient sampling technique will be used to recruit the individuals into two groups. Group A had undergone Senobi exercises and Group B engaged in Jacobsons Muscular relaxation exercises along with conventional treatment of COPD.

DETAILED DESCRIPTION:
It will be a randomized clinical trial with 40 participants, aimed to compare the effects of Senobi and Jacobsons muscular relaxation exercises on pulmonary functions, dyspnea, and sleep quality in COPD patients. Participants were chosen through convenient sampling at Sarwet Anver Medical Complex Lahore. Participants were divided into Groups A and B. Group A had undergone Senobi exercises and Group B had engaged in Jacobsons muscular relaxation exercises. The pulmonary function was assessed by spirometer the calculated values will be FVC (Forced vital capacity) and FEV1(Forced expiratory volume in one second). The dyspnea will be assessed by a 6-minute walk test and at the end of the walk state of breathlessness will be evaluated by the Modified Borg Dyspnea Scale. The sleep quality will be assessed by the SATED sleep questionnaire The exercises were evaluated after 6 weeks of interventions. Data was analyzed using SPSS software version 2.5.

Spirometry assesses the amount and speed of air that can be inhaled and exhaled. Key measurements include Forced Vital Capacity (FVC). The maximum volume of air forcefully exhaled after a full inhalation. Forced Expiratory Volume in 1 second (FEV1): The volume of air exhaled in the first second of the FVC test, indicates how quickly the lungs can be emptied.

The modified Borg dyspnea score is a variation of the CR10 scale, with a range from 0 to 10, where 0 signifies the absence of breathlessness and 10 indicates the highest level of breathlessness. Participants assess their dyspnea after the 6-minute walk distance (6MWD) test, capturing the peak intensity of breathlessness experienced throughout the entire walking test. This scoring system provides a subjective measure of the individual's maximal perceived dyspnea during physical activity.

The SATED scale includes specific quantitative criteria for four of the five sleep-related dimensions that have been reliably linked to health outcomes. It evaluates five important aspects of sleep. These include the following dimensions: sleep satisfaction, sleep efficiency, sleep duration, timing of sleep, and alertness during waking hours.

ELIGIBILITY:
Inclusion Criteria:

Both genders

* Age 35-50 years
* Diagnosed COPD patients of stage 2-3 according to gold criteria (moderate)

Exclusion Criteria:

* Patients with neurological disorders
* History of fractures (68)
* History of other pulmonary complications

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-10-25 (Estimated)

PRIMARY OUTCOMES:
FEV1(Forced Expiratory Volume per second) | Pre and Post after 6 week
  Pulmonary Function Test using Digital Spirometer
FVC(Forced Vital Capacity) | Pre and Post after 6 week
  Pulmonary Function Test using Digital Spirometer
Modified Borg dyspnea Scale | Pre and Post after 6 week
  To asses dyspnea
6-minutes walk Test | Pre and Post after 6 week
  To asses dyspnea
SATED SLEEP questionnaire | Pre and Post after 6 week
  To asses sleep

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Shehzadi, Mphil, Principal Investigator — Riphah International University
Locations (1):
- University of Lahore Teaching Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No